CLINICAL TRIAL: NCT02760433
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled, Multicenter Phase III Study of the Efficacy and Safety of Olokizumab in Subjects With Moderately to Severely Active Rheumatoid Arthritis Inadequately Controlled by Tumor Necrosis Factor Alpha (TNF-α) Inhibitor Therapy
Brief Title: Evaluation of the Efficacy and Safety of Two Dosing Regimens of Olokizumab (OKZ), Compared to Placebo, in Subjects With Rheumatoid Arthritis (RA) Who Were Taking an Existing Medication Called a Tumour Necrosis Factor Alpha Inhibitor But Had Active Disease
Acronym: CREDO 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: Quintiles, Inc. (Industry); OCT Clinical Trials (Other); Mene Research (Other)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL04041025; 2015-005308-27 (EudraCT Number)
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Results first posted 2021-07-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
Keywords: moderate Rheumatoid Arthritis; severe Rheumatoid Arthritis; Olokizumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — olokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Olokizumab q4w (Experimental): Olokizumab 64mg subcutaneous q4w + placebo + Methotrexate
  Olokizumab 64 mg subcutaneous q4w + placebo+ concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular) in order to maintain the blind, subjects randomized to receive OKZ q4w received placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.)
  Interventions: Drug: Olokizumab; Drug: Placebo
- Arm 2: Olokizumab q2w (Experimental): Olokizumab 64mg subcutaneous q2w + Methotrexate
  64 mg Olokizumab administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
  Interventions: Drug: Olokizumab
- Arm 3: Placebo q2w (Placebo Comparator): Placebo q2w subcutaneous + Methotrexate
  Placebo administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
  Starting at Week 16, all subjects in the placebo group were randomized in a blinded fashion to receive either OKZ 64 mg q2w or OKZ 64 mg q4w; equal numbers of subjects were planned to be assigned to each OKZ treatment group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olokizumab — 160 mg/mL sterile solution for SC injection in a 2 mL clear Type I glass vial
  Arms: Arm 1: Olokizumab q4w; Arm 2: Olokizumab q2w
Drug: Placebo — sodium chloride 0.9% solution provided as either a 10 mL vial or ampoule, depending on market availability. Each placebo will be packed into a cardboard carton to contain 1 vial or ampoule
  Arms: Arm 1: Olokizumab q4w; Arm 3: Placebo q2w

SUMMARY:
The purpose of this study was to determine how effective and safe the study drug Olokizumab was in patients with Rheumatoid Arthritis (RA) who had been already receiving, but not fully responding to treatment with an existing medication called a tumour necrosis factor alpha inhibitor

The primary objective of this study was to evaluate the efficacy of olokizumab (OKZ) 64 mg administered subcutaneously (SC) once every 2 weeks (q2w) or once every 4 weeks (q4w) relative to placebo in subjects with moderately to severely active rheumatoid arthritis (RA) inadequately controlled by TNF-α inhibitor (TNFi) therapy.

DETAILED DESCRIPTION:
The goal of this Phase III study was to assess the efficacy, safety and tolerability of OKZ in subjects with moderately to severely active RA who had responded inadequately to TNFi therapy. The primary endpoint of the trial was assessed at Week 12. Olokizumab was expected to reduce the disease activity and improve physical function. The study was expected to provide safety information in a large group of subjects over at least a 24 week period.

This was a randomized, double-blind, parallel-group, placebo-controlled, multicenter study. This study included a 4-week Screening Period, a double-blind Treatment Period from Week 0 to Week 24, and a Safety FollowUp Period from Week 24 to Week 44.

A total of 350 subjects were planned to be randomized.Subjects were assessed for eligibility to enter the study during a 4-week Screening Period. Eligible subjects were randomized at Visit 2 in a 2:2:1 ratio in one of 3 treatment groups (planned 140, 140, and 70 subjects per group, respectively) :

1. Olokizumab 64 mg q4w: SC injection of OKZ 64 mg q4w (alternating with SC injection of placebo OKZ q4w to maintain blinding) + MTX for 24 weeks,
2. Olokizumab 64 mg q2w: SC injection of OKZ 64 mg q2w + MTX for 24 weeks or
3. Placebo: SC injection of placebo q2w + MTX for 16 weeks.

Subjects who received placebo were re-randomized at Week 16 to receive 64 mg OKZ q4w + Methotrexate or 64 mg OKZ q2w +Methotrexate for 8 weeks.

Throughout the double-blind Treatment Period, all subjects were required to remain on a stable dose of background MTX with a stable route of administration. Concomitant treatment with folic acid was required for all subjects. The last dose of OKZ was administered at Week 20 for subjects receiving OKZ 64 mg q4w and at Week 22 for subjects receiving OKZ 64 mg q2w.

Following Visit 2 (randomization; Week 0), subjects returned to the study site at least every 2 weeks through Week 24 for response and safety assessments.

At Week 14, subjects who did not improve by at least 20% in both swollen and tender joint counts were classified as nonresponders and were administered sulfasalazine and/or hydroxychloroquine as rescue medication in addition to the assigned treatment.

After completion of the 24-week double-blind Treatment Period, subjects either rolled over into the long-term open-label extension (OLE) study or entered the Safety Follow-Up Period. During the Safety Follow-Up Period, subjects returned for visits +4, +8, and +22 weeks after the last dose of study treatment.

Subjects who discontinued randomized treatment prematurely were required to come for the End of Treatment (EoT) Visit 2 weeks after the last study treatment administration and then continue with the scheduled study visits.

Adverse events (AEs) were assessed throughout the study (starting when the subject signed the informed consent form) and evaluated using the Common Terminology Criteria for Adverse Events Version 4.0. There was ongoing monitoring of safety events, including laboratory findings, by the Sponsor or the Sponsor's designee. In addition, safety was assessed throughout the study by an independent Data Safety Monitoring Board and potential major adverse cardiac events were evaluated by an independent Cardiovascular Adjudication Committee.

The study was conducted at 123 sites across 11 countries globally (in US,EU, Russian Federation, Asia, Latin America)

ELIGIBILITY:
Inclusion Criteria:

Subjects may be enrolled in the study only if they meet all of the following criteria.

* Subjects willing and able to sign informed consent
* Subjects must have a diagnosis of adult onset RA classified by ACR/EULAR 2010 revised classification criteria for RA for at least 24 weeks prior to Screening.

(If the subject was diagnosed according to ACR 1987 criteria previously, the Investigator may classify the subject per ACR 2010 retrospectively, using available source data.)

* Treatment with oral, SC, or intramuscular (IM) MTX for at least 12 weeks prior to Screening at a dose of 15 to 25 mg/week (or ≥10 mg/week if there is documented intolerance to higher doses)

  * The dose and means of administering MTX must have been stable for at least 6 weeks prior to Screening.
* Subjects must be willing to take folic acid or equivalent throughout the study.
* Subjects must have moderately to severely active RA disease as defined by all of the following:

  * ≥6 tender joints (68 joint count) at Screening and baseline; and
  * ≥6 swollen joints (66 joint count) at Screening and baseline; and
  * C-reactive protein (CRP) above Upper limit of normal (ULN) at Screening based on the central laboratory results.
* Subjects must have a documented inadequate response to treatment (i.e., TNFi failure) with ≥1 licensed TNFi following at least 12 weeks of therapy with that agent. Inadequate response to treatment is classified as either:

  * Primary failure: The absence of any documented clinically significant response; or
  * Secondary failure: Documented initial response with subsequent loss of that response or partial response

Exclusion Criteria:

* Diagnosis of any other inflammatory arthritis or systemic rheumatic disease (e.g., gout, psoriatic or reactive arthritis, Crohn's disease, Lyme disease, juvenile idiopathic arthritis, or systemic lupus erythematosus) (However, subjects may have secondary Sjogren's syndrome or hypothyroidism.)
* Subjects who are Steinbrocker class IV functional capacity (incapacitated, largely or wholly bed-ridden or confined to a wheelchair, with little or no self-care)
* Prior exposure to any licensed or investigational compound directly or indirectly targeting Interleukin (IL) 6 or IL 6R (including tofacitinib or other Janus kinases and spleen tyrosine kinase [SYK] inhibitors)
* Prior treatment with cell depleting therapies including anti CD20 or investigational agents (e.g., CAMPATH, anti CD4, anti CD5, anti CD3, and anti CD19) with the exception of rituximab, which is allowed if it was discontinued at least 24 weeks prior to baseline (rituximab should not be discontinued to facilitate a subject's participation in the study, but should instead have been previously discontinued as part of a subject's medical management of RA).
* Prior use of bDMARDs, within the following windows prior to baseline (bDMARDs should not be discontinued to facilitate a subject's participation in the study, but should instead have been previously discontinued as part of a subject's medical management of RA):

  1. 4 weeks for etanercept and anakinra
  2. 8 weeks for infliximab
  3. 10 weeks for adalimumab, certolizumab, and golimumab
  4. 12 weeks for abatacept
* Use of parenteral and/or intra-articular glucocorticoids within 4 weeks prior to baseline
* Use of oral glucocorticoids greater than 10 mg/day prednisone (or equivalent) or change in dosage within 2 weeks prior to baseline
* Prior documented history of no response to hydroxychloroquine and sulfasalazine
* Prior use of cDMARDs (other than MTX) within the following windows prior to baseline (cDMARDs should not be discontinued to facilitate a subject's participation in the study, but should instead have been previously discontinued as part of a subject's medical management of RA):

  1. 4 weeks for sulfasalazine, azathioprine, cyclosporine, hydroxychloroquine, chloroquine, gold, penicillamine, minocycline, or doxycycline
  2. 12 weeks for leflunomide unless the subject has completed the following elimination procedure at least 4 weeks prior to baseline: Cholestyramine at a dosage of 8 grams 3 times daily for at least 24 hours, or activated charcoal at a dosage of 50 grams 4 times daily for at least 24 hours
  3. 24 weeks for cyclophosphamide
* Vaccination with live vaccines in the 6 weeks prior to baseline or planned vaccination with live vaccines during the study
* Participation in any other investigational drug study within 30 days or 5 times the terminal half-life of the investigational drug, whichever is longer, prior to baseline
* Other treatments for RA (e.g., Prosorba Device/Column) within 6 months prior to baseline
* Use of intra-articular hyaluronic acid injections within 4 weeks prior to baseline
* Use of non steroidal anti inflammatory drugs (NSAIDs) on unstable dose or switching of NSAIDs within 2 weeks prior to baseline
* Previous participation in this study (randomized) or another study of OKZ
* Subjects with concurrent acute or chronic viral Hepatitis B or C infection as detected by blood tests at Screening (e.g., positive for hepatitis B surface antigen [HBsAg], total hepatitis B core antibody [anti-HBc], or hepatitis C virus antibody [HCV Ab])

  a) subjects who are positive for hepatitis B surface antibodies (anti-HBs), but negative for HBsAg and anti-HBc, will be eligible.
* Subjects with HIV infection
* Subjects with:

  1. Suspected or confirmed current active tuberculosis (TB) disease or a history of active TB disease.
  2. Close contact (i.e., sharing the same household or other enclosed environment, such as a social gathering place, workplace, or facility, for extended periods during the day) with an individual with active TB within 1.5 years prior to Screening
* Concurrent malignancy or a history of malignancy within the last 5 years (with the exception of successfully treated carcinoma of the cervix in situ and successfully treated basal cell carcinoma and squamous cell carcinoma not less than 1 year prior to Screening [and no more than 3 excised skin cancers within the last 5 years prior to Screening])
* Subjects with any infection requiring oral antibiotic or antiviral therapy in the 2 weeks prior to Screening or at baseline, injectable anti-infective therapy in the last 4 weeks prior to baseline, or serious or recurrent infection with history of hospitalization in the 6 months prior to baseline
* Subjects with evidence of disseminated herpes zoster infection, zoster encephalitis, meningitis, or other non-self-limited herpes zoster infections in the 6 months prior to baseline
* Subjects with planned surgery during the study or surgery ≤ 4 weeks prior to Screening and from which the subject has not fully recovered, as judged by the Investigator
* Subjects with diverticulitis or other symptomatic GI conditions that might predispose the subject to perforations, including subjects with history of such predisposing conditions (e.g., diverticulitis, GI perforation, or ulcerative colitis)
* Pre-existing central nervous system demyelinating disorders (e.g., multiple sclerosis and optic neuritis)
* History of chronic alcohol or drug abuse as judged by the Investigator
* Subjects with a known hypersensitivity to any component of the OKZ drug product or placebo
* Subjects with a known hypersensitivity or contraindication to any component of the rescue medication
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Female subjects who are pregnant, currently lactating, have lactated within the last 12 weeks, or who are planning to become pregnant during the study or within 6 months of the last dose of study treatment
* Female subjects of childbearing potential (unless permanent cessation of menstrual periods, determined retrospectively after a woman has experienced 12 months of natural amenorrhea as defined by the amenorrhea with underlying status [e.g., correlative age] or 6 months of natural amenorrhea with documented serum follicle-stimulating hormone levels >40 mIU/mL and estradiol <20 pg/mL) who are not willing to use a highly effective method of contraception during the study and for at least 6 months after the last administration of study treatment

OR

Male subjects with partners of childbearing potential not willing to use a highly effective method of contraception during the study and for at least 3 months after the last administration of study treatment.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (116):
- United States (50):
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - CHI St. Vincent Hot Springs, Hot Springs, Arkansas
  - Medvin Clinical Research, Covina, California
  - TriWest Research Associates, LLC, El Cajon, California
  - Saint Jude Heritage Medical Grp, Fullerton, California
  - С V Mehta MD Med Corp., Hemet, California
  - Advanced Medical Research, LLC, Lakewood, California
  - Stanford University School of Medicine, Palo Alto, California
  - Riverside Medical Clinic, Riverside, California
  - East Bay Rheumatology Medical Group, Inc., San Leandro, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Javed Rheumatology Associates, Newark, Delaware
  - RASF - Clinical Research Center, Boca Raton, Florida
  - Suncoast Research Group LLC, Miami, Florida
  - Omega Research Consultants, Orlando, Florida
  - Family Clinical Trials, LLC., Pembroke Pines, Florida
  - AdventHealth Medical Group, PA, Tampa, Florida
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - University of Kansas Hospital, Kansas City, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - The Arthritis & Diabetes Clinic, Inc., Monroe, Louisiana
  - Klein and Associates, M.D., P.A., Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Glacier View Research Instutute-Rheumatology, Kalispell, Montana
  - Arthritis & Osteoporosis Associates, PA, Freehold, New Jersey
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - NYU Langone Ambulatory Care, New York, New York
  - Medication Management, LLC, Greensboro, North Carolina
  - Cape Fear Arthritis Care, Leland, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - Trinity Medical Group, Minot, North Dakota
  - Cincinnati Rheumatic Disease Study Group, Cincinnati, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - Clinical Research Source, Inc., Perrysburg, Ohio
  - Arthritis Group, Philadelphia, Pennsylvania
  - Low Country Research Center, Charleston, South Carolina
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Austin Regional Clinic, P.A., Austin, Texas
  - Accurate Clinical Research, Inc., Baytown, Texas
  - Precision Comprehensive Clinical Research Solutions, Grapevine, Texas
  - Therapeutic Concepts Rheumatology, LLC, Houston, Texas
  - Rheumatology Clinic of Houston, P.A., Houston, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Accurate Clinical Research, Inc., League City, Texas
  - Endocrinology, Internal Medicine, Lubbock, Texas
  - Dr. Alex De Jesus Rheumatology, P.A., San Antonio, Texas
  - Advanced Rheumatology of Houston, Woodville, Texas
- Argentina (13):
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Clinica de Higado y Aparato Digestivo, Rosario, Santa Fe Province
  - Sanatorio San Martin, Venado Tuerto, Santa Fe Province
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán, Tucumán Province
  - Atencion Integral en Reumatologia (AIR), Ciudad Autonoma Buenos Aires
  - Organizacion Medica de Investigacion (OMI), Ciudad Autonoma Buenos Aires
  - APRILLUS, Ciudad Autonoma Buenos Aires
  - Instituto Centenario, Ciudad Autonoma Buenos Aires
  - Hospital Privado Centro Medico de Cordoba S.A, Córdoba
  - Centro Polivalente de Asistencia e Inv. Clinica CER, San Juan
- Brazil (12):
  - HUWC - UFC - Hospital Universitário Walter Cantídio - Universidade Federal do Ceará, Fortaleza, Ceará
  - CEDOES - Diagnóstico e Pesquisa, Vitória, Espírito Santo
  - CIP - Centro Internacional de Pesquisa, Goiânia, Goiás
  - CMiP - Centro Mineiro de Pesquisa, Juiz de Fora, Minas Gerais
  - CETI - Centro de Estudos em Terapias Inovadoras Ltda., Curitiba, Paraná
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - LMK Serviços Médicos S/S Ltda, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos - CEMEC, São Bernardo do Campo, São Paulo
  - Clínica de Neoplasias Litoral Ltda., Santa Catarina
  - CPCLIN - Centro de Pesquisas Clínicas Ltda., São Paulo
  - Associação de Assistência à Criança Deficiente - AACD, São Paulo
- Colombia (4):
  - Centro de Reumatologia y Ortopedia SAS, Barranquilla
  - Centro de Investigacion en Reumatologia y Especialidades Medicas SAS. CIREEM, Bogotá
  - Medicity S.A.S., Bucaramanga
  - Clinica de Artritis Temprana S.A., Cali
- Czechia (4):
  - Revmatologie MUDr. Klara Sirova s.r.o., Ostrava - Moravska Ostrava
  - CCR Czech, a.s., Pardubice
  - MEDICAL PLUS s.r.o., Uherské Hradiště
  - PV - Medical, s.r.o., Zlín
- Germany (3):
  - Kerckhoff-Klinik gGmbH, Bad Nauheim, Hesse
  - SMO.MD GmbH, Magdeburg, Saxony-Anhalt
  - HRF Hamburger Rheuma Forschungszentrum, Hamburg
- Hungary (4):
  - Clinexpert Egeszsegugyi Szolg. es Ker. Kft., Budapest
  - Obudai Egeszsegugyi Centrum, Budapest
  - MAV Korhaz és Rendelointezet, Szolnok
  - Vital Medical Center, Veszprém
- Mexico (8):
  - Clinica de Investigacion en Reumatologia y Obesidad S.C., Guadalajara, Jalisco
  - Centro de Estudios de Investigacion Basica y Clinica SC, Guadalajara, Jalisco
  - Centro de Investigacion Clínica GRAMEL S.C, Mexico City, Mexico City
  - Clinstile, S.A. de C.V., Mexico City, Mexico City
  - Accelerium S. de R.L. de C.V., Monterrey, Nuevo León
  - Universidad Autonoma de Nuevo Leon, Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Centro de Alta Especialidad en Reumatología e Investigación del Potosí, S.C., San Luis Potosí City, San Luis Potos
  - Investigacion y Biomedicina de Chihuahua, S.C., Chihuahua City
- Poland (6):
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - McBk S.C., Grodzisk Mazowiecki
  - Centrum Medyczne AMED, Lodz
  - Szpital Wojewodzki im. Prymasa Kardynala Stefana Wyszynskiego, Sieradz
  - Samodzielny Publiczny ZOZ Tomaszow Lubelski, Tomaszów Lubelski
  - McM Polimedica, Warsaw
- Russia (8):
  - State Budgetary Healthcare Institution "City Clinical Hospital # 15 n.a O.M. Filatov" of Moscow Healtheare Department, Moscow, Moscow Oblast
  - City Clinical Hospital #1, Novosibirsk, Novosibirsk Oblast
  - Diagnostic Center Ultramed, Omsk, Omsk Oblast
  - SBHI of the Republic of Karelia "Republican Hospital named after V.A.Baranov", Petrozavodsk, Republic of Karelia
  - Rostov State Medical Unversity, Rostov-on-Don, Rostov Oblast
  - SBHI of Stavropol Region "Stavropol Regional Clinical Hospital", Stavropol, Stavropol Kray
  - Regional Clinical Hospital, Vladimir, Vladimirskaya Oblast’
  - FSBSI "Scientific Research Institute of Rheumatology n.a. V.A. Nasonova", Moscow
- South Korea (4):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chonnam National University Hospital, Gwangju
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Severance Hospital, Yonsei University, Seoul

REFERENCES:
- [Derived] Feist E, Fatenejad S, Grishin S, Korneva E, Luggen ME, Nasonov E, Samsonov M, Smolen JS, Fleischmann RM. Olokizumab, a monoclonal antibody against interleukin-6, in combination with methotrexate in patients with rheumatoid arthritis inadequately controlled by tumour necrosis factor inhibitor therapy: efficacy and safety results of a randomised controlled phase III study. Ann Rheum Dis. 2022 Dec;81(12):1661-1668. doi: 10.1136/ard-2022-222630. Epub 2022 Sep 15. PMID 36109142

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 123 clinical sites across 11 countries (US,EU, Russian Federation, Asia, Latin America). 718 subjects were screened and 368 subjects were enrolled (randomized) and treated, 318 subjects completed the study. A total of 368 subjects were analyzed for efficacy in the ITT Population and 368 subjects were analyzed for safety in the Safety Population.
Groups:
- Arm 1: Olokizumab q4w: Olokizumab 64mg subcutaneous q4w +placebo + Methotrexate
  Olokizumab 64 mg subcutaneous q4w + placebo+ concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular) in order to maintain the blind, subjects randomized to receive OKZ q4w received placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.)
  There was no re-randomization at week 16 for this arm
- Arm 2: Olokizumab q2w: Olokizumab 64mg subcutaneous q2w + Methotrexate
  64 mg Olokizumab administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
  There was no re-randomization at week 16 for this arm
- Arm 4: Placebo-OKZ 64 mg q4w: refers to subjects who initially received placebo q2w (Arm 3: Placebo administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate), but then were re-randomized at week 16 to receive OKZ 64 mg q4w. Arm 3 (placebo q2w) consisted of subjects from arms 4, 5 and 8).
  (Arm 6 (Any Olokizumab q4w) combines the subjects from Arm 1 and Arm 4 (AEs were collected starting from the first OKZ dose after rerandomization). This group is included in the safety data presentation).
- Arm 5: Placebo-OKZ 64 mg q2w: refers to subjects who initially received placebo q2w (Arm 3:Placebo administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate), but then were re-randomized at week 16 to receive OKZ 64 mg q2w. Arm 3 (placebo q2w) consisted of subjects from arms 4, 5 and 8).
  (Arm 7 (Any Olokizumab q2w) combines the subjects from Arm 2 and Arm 5 (AEs were collected starting from the first OKZ dose after rerandomization). This group is included in the safety data presentation).
- Arm 8: Placebo Only: refers to subjects who were initially randomized to placebo q2w (Arm3: Placebo administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate), but who were not re-randomized to OKZ 64 mg q2w or OKZ 64 mg q4w. Arm 3 (placebo q2w) consisted of subjects from arms 4, 5 and 8).
Period: Overall Study
Arm/Group | Arm 1: Olokizumab q4w | Arm 2: Olokizumab q2w | Arm 4: Placebo-OKZ 64 mg q4w | Arm 5: Placebo-OKZ 64 mg q2w | Arm 8: Placebo Only
Started | 161 | 138 | 26 | 32 | 11
Completed | 134 | 128 | 25 | 30 | 1
Not Completed | 27 | 10 | 1 | 2 | 10
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 23 | 9 | 0 | 2 | 9
Not completed — Lack of Response At Week 14 | 0 | 0 | 0 | 0 | 1
Not completed — Subject refused to continue the study | 1 | 0 | 0 | 0 | 0
Not completed — Subject was taking prohibited medications and refused to stop. | 2 | 0 | 0 | 0 | 0
Not completed — Ongoing Adverse Events (low platelet count) with long interruptions of investigational product | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Arm 3 (Placebo) combines all subjects from Arms 4, 5 and 8. Starting at Week 16, subjects in the placebo group were randomized in a blinded fashion to receive either OKZ 64 mg q2w or OKZ 64 mg q4w. (Efficacy data are presented for Arm 1, Arm 2, and Arm 3.)
Groups:
- Arm 1: Olokizumab q4w: Olokizumab 64mg subcutaneous q4w +placebo + Methotrexate
  Olokizumab 64 mg subcutaneous q4w + placebo+ concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular) in order to maintain the blind, subjects randomized to receive OKZ q4w received placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.)
- Arm 4: Placebo-OKZ 64 mg q4w: refers to subjects who initially received placebo q2w, but then were re-randomized at week 16 to receive OKZ 64 mg q4w
  (Arm 6 (Any Olokizumab q4w) combines the subjects from Arm 1 and Arm 4 (AEs were collected starting from the first OKZ dose after rerandomization). This group is included in the safety data presentation.)
- Arm 5: Placebo-OKZ 64 mg q2w: refers to subjects who initially received placebo q2w, but then were re-randomized at week 16 to receive OKZ 64 mg q2w
  (Arm 7 (Any Olokizumab q2w) combines the subjects from Arm 2 and Arm 5 (AEs were collected starting from the first OKZ dose after rerandomization). This group is included in the safety data presentation.)
- Arm 8: Placebo Only: refers to subjects who were initially randomized to placebo, but who were not re-randomized to OKZ 64 mg q2w or OKZ 64 mg q4w
- Total: Total of all reporting groups
Arm/Group | Arm 1: Olokizumab q4w | Arm 2: Olokizumab q2w | Arm 4: Placebo-OKZ 64 mg q4w | Arm 5: Placebo-OKZ 64 mg q2w | Arm 8: Placebo Only | Total
Number analyzed (Participants) | 161 | 138 | 26 | 32 | 11 | 368
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 132 | 114 | 20 | 27 | 7 | 300
  >=65 years | 29 | 24 | 6 | 5 | 4 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (11.68) | 53.4 (12.68) | 53.5 (14.13) | 53.9 (11.67) | 48.9 (18.28) | 53.5 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 122 | 20 | 27 | 8 | 307
  Male | 31 | 16 | 6 | 5 | 3 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 6 | 1 | 1 | 0 | 11
  Black of African American | 11 | 11 | 0 | 1 | 0 | 23
  White | 139 | 110 | 19 | 24 | 10 | 302
  Other/Mixed | 8 | 11 | 6 | 6 | 1 | 32
Region of Enrollment [Number; unit: participants]
  Colombia | 3 | 5 | 2 | 3 | 0 | 13
  Argentina | 14 | 11 | 1 | 2 | 0 | 28
  South Korea | 1 | 2 | 0 | 1 | 0 | 4
  Hungary | 8 | 10 | 2 | 3 | 1 | 24
  United States | 63 | 44 | 10 | 8 | 3 | 128
  Czechia | 17 | 13 | 2 | 2 | 2 | 36
  Brazil | 8 | 11 | 1 | 3 | 1 | 24
  Poland | 5 | 5 | 0 | 2 | 1 | 13
  Mexico | 27 | 28 | 8 | 8 | 2 | 73
  Germany | 3 | 1 | 0 | 0 | 0 | 4
  Russia | 12 | 8 | 0 | 0 | 1 | 21
Body Mass Index (BMI),Continuous [Mean (Full Range); unit: kg/m^2] | 29.218 [17.99 to 56.25] | 28.755 [17.78 to 57.93] | 28.895 [20.74 to 49.93] | 28.467 [17.82 to 37.60] | 26.976 [21.09 to 38.37] | 28.888 [17.78 to 57.93]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving American College of Rheumatology 20% (ACR20) Response
Description: The difference between OKZ and placebo in the percentage of subjects achieving an ACR20 response and remaining on randomized treatment and in the study at Week 12. A responder is defined as any subject satisfying ACR20 criteria and remaining on randomized treatment and in the study at Week 12.
  American College of Rheumatology 20 % response is a composite defined as a ≥ 20% improvement from baseline in the swollen joint counts assessed in 66 joints and in the tender joint count assessed in 68 joints; and a ≥20% improvement from baseline in at least 3 of the 5 remaining core set measures:
  * Patient Global Assessment of Disease Activity (VAS)
  * Patient Assessment of Pain (VAS)
  * HAQ-DI
  * Physician Global Assessment (VAS)
  * Level of acute phase reactant (CRP)
Time Frame: at Week 12
Population: Intent-to-treat (ITT) population: The ITT population includes all randomized subjects. Subjects were analyzed according to the treatment group to which they were randomized. The ITT population is the primary analysis population.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Olokizumab 64 mg q4w: Olokizumab 64mg subcutaneous q4w +placebo + Methotrexate
  Olokizumab 64 mg subcutaneous q4w + placebo+ concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular) in order to maintain the blind, subjects randomized to receive OKZ q4w received placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.)
- Arm 2: Olokizumab 64 mg q2w: Olokizumab 64mg subcutaneous q2w + Methotrexate
  64 mg Olokizumab administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
- Arm 3: Placebo q2w: Placebo q2w subcutaneous + Methotrexate
  Placebo administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
  Starting at Week 16, all subjects in the placebo group were randomized in a blinded fashion to receive either OKZ 64 mg q2w or OKZ 64 mg q4w;
  Arm 3 (placebo q2w) consisted of subjects from arms 4, 5 and 8 reported previously
Arm/Group | Arm 1: Olokizumab 64 mg q4w | Arm 2: Olokizumab 64 mg q2w | Arm 3: Placebo q2w
Number analyzed (Participants) | 161 | 138 | 69
Participants | 96 | 84 | 28
Statistical Analysis 1: Comparison: Arm 1: Olokizumab 64 mg q4w vs Arm 3: Placebo q2w; The ACR20 response rate at Week 12 for the placebo group is estimated to be 20% in this study population. The OKZ ACR20 response rate for 64 mg q4w treatment group at Week 12 are expected to be at least 45%, resulting in an expected difference in ACR20 response rates of 25 percentage points between the respective OKZ treatment group and placebo. Sample size yield 100% disjunctive power for testing the primary hypothesis; Test type: Superiority; p = 0.004, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.190, 97.5% CI 2-sided [0.030 to 0.337]
Statistical Analysis 2: Comparison: Arm 2: Olokizumab 64 mg q2w vs Arm 3: Placebo q2w; The ACR20 response rate at Week 12 for the placebo group is estimated to be 20% in this study population .The OKZ ACR20 response rate for 64 mg q2w treatment group at Week 12 is expected to be at least 50%, resulting in an expected difference in ACR20 response rates of 30 percentage points between the respective OKZ treatment group and placebo. Sample size yield 100% disjunctive power for testing the primary hypothesis; Test type: Superiority; p = 0.0029, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.203, 97.5% CI 2-sided [0.038 to 0.353]

2. Secondary Outcome: Percentage of Subjects Achieving Low Disease Activity
Description: Defined as Disease Activity Score 28-joint count (DAS28) C-reactive protein (CRP) <3.2, and remaining on randomized treatment and in the study at Week 12
Time Frame: at Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Olokizumab q4w | Arm 2: Olokizumab q2w | Arm 3: Placebo q2w
Number analyzed (Participants) | 161 | 138 | 69
Participants | 47 | 55 | 8
Statistical Analysis 1: Comparison: Arm 1: Olokizumab q4w vs Arm 3: Placebo q2w; The DAS28 low disease activity (based on DAS28 [CRP] <3.2) response rate at Week 12 was estimated to be 5% in the placebo group and 18% and 21% in 64 mg q4w and q2w OKZ groups, respectively, resulting in an expected difference of 13 and 16 percentage points between respective OKZ groups and placebo; Test type: Superiority; p = 0.0021, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.176, 97.5% CI 2-sided [0.041 to 0.281]
Statistical Analysis 2: Comparison: Arm 2: Olokizumab q2w vs Arm 3: Placebo q2w; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.283, 97.5% CI 2-sided [0.139 to 0.396]

3. Secondary Outcome: Improvement of Physical Ability From Baseline to Week 12, as Measured by the Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: Change of physical ability from baseline (the last available assessment prior to the first dose of the study treatment) to week 12, as measured by HAQ-DI. The HAQ-DI assesses the degree of difficulty experienced in 8 domains of daily living activities using 20 questions.The domains are dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities, and each domain consists of 2 or 3 items. For each question, the level of difficulty is scored from 0 to 3 where 0 = without any difficulty (the best outcome), 1 = with some difficulty, 2 = much difficulty, and 3 = unable to do (the worst outcome). Each category is given a score by taking the maximum score of each question. A decrease from baseline indicates improvement for HAQ-DI.The HAQ-DI was calculated by dividing the sum of the category scores by the number of categories with at least 1 question answered. The HAQ-DI total score ranges from 0 (the best outcome) to 3 (the worst outcome).
Time Frame: Baseline to Week 12
Population: Intent-to-treat (ITT) population: The ITT population includes all randomized subjects. Subjects were analyzed according to the treatment group to which they were randomized. The ITT population is the primary analysis population. Subjects with a missing baseline are not included. Data after treatment discontinuation are Included, Data after discontinuing study are multiply Imputed based on the return to baseline assumption.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: Olokizumab q4w | Arm 2: Olokizumab q2w | Arm 3: Placebo q2w
Number analyzed (Participants) | 157 | 131 | 68
score on a scale | -0.39 (0.048) | -0.49 (0.056) | -0.32 (0.063)
Statistical Analysis 1: Comparison: Arm 1: Olokizumab q4w vs Arm 3: Placebo q2w; Test type: Superiority; p = 0.1814, ANCOVA — p-value was greater than the threshold p-value of 0.0125; Least Squares Mean Difference = -0.07, 97.5% CI 2-sided [-0.26 to 0.11], Standard Error of Mean 0.081
Statistical Analysis 2: Comparison: Arm 2: Olokizumab q2w vs Arm 3: Placebo q2w; Test type: Superiority; p = 0.0227, ANCOVA — p-value was greater than the threshold p-value of 0.0125; Least Squares Mean Difference = -0.17, 97.5% CI 2-sided [-0.35 to 0.02], Standard Error of Mean 0.083

4. Secondary Outcome: Percentage of Subjects Achieving American College of Rheumatology 50% (ACR50) Response
Description: Difference between OKZ and placebo in the percentage of subjects achieving an ACR50 response and remaining on randomized treatment and in the study at Week 12.
  American College of Rheumatology 50% Response is a composite defined as ≥50%, improvement from baseline in the swollen joint counts assessed in 66 joints and in the tender joint count assessed in 68 joints; and a ≥50%, improvement from baseline in at least 3 of the 5 remaining core set measures:
  * Patient Global Assessment of Disease Activity (VAS)
  * Patient Assessment of Pain (VAS)
  * HAQ-DI
  * Physician Global Assessment (VAS)
  * Level of acute phase reactant (CRP)
Time Frame: at Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Arm 3: Placebo q2w: Placebo q2w subcutaneous + Methotrexate
  Placebo q2w subcutaneous + Methotrexate
  Placebo administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
  Starting at Week 16, all subjects in the placebo group were randomized in a blinded fashion to receive either OKZ 64 mg q2w or OKZ 64 mg q4w;
  Arm 3 (placebo q2w) consisted of subjects from arms 4, 5 and 8 reported previously
Arm/Group | Arm 1: Olokizumab q4w | Arm 2: Olokizumab q2w | Arm 3: Placebo q2w
Number analyzed (Participants) | 161 | 138 | 69
Participants | 52 | 46 | 11
Statistical Analysis 1: Comparison: Arm 1: Olokizumab q4w vs Arm 3: Placebo q2w; Test type: Superiority; Due to the hierarchical nature of pre-planned statistical testing (gate-keeping strategy) a formal statement could not be made; Risk Difference (RD) = 0.164, 97.5% CI 2-sided [0.020 to 0.278]
Statistical Analysis 2: Comparison: Arm 2: Olokizumab q2w vs Arm 3: Placebo q2w; Test type: Superiority; [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = 0.174, 97.5% CI 2-sided [0.027 to 0.294]

5. Secondary Outcome: Percentage of Subjects With Clinical Disease Activity Index (CDAI) ≤ 2.8 (Remission)
Description: Difference between OKZ and placebo in the percentage of subjects with Clinical Disease Activity Index (CDAI) ≤2.8 (remission) and remaining on randomized treatment and in the study at Week 12
Time Frame: at Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Olokizumab q4w | Arm 2: Olokizumab q2w | Arm 3: Placebo q2w
Number analyzed (Participants) | 161 | 138 | 69
Participants | 5 | 9 | 0
Statistical Analysis 1: Comparison: Arm 1: Olokizumab q4w vs Arm 3: Placebo q2w; Test type: Superiority; [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = 0.031, 97.5% CI 2-sided [-0.052 to 0.083] — means continuity correction applied because expected cell counts < 5
Statistical Analysis 2: Comparison: Arm 2: Olokizumab q2w vs Arm 3: Placebo q2w; Test type: Superiority; [p-value comment as in outcome 4, analysis 1]; Risk Difference (RD) = 0.065, 97.5% CI 2-sided [-0.023 to 0.134] — means continuity correction applied because expected cell counts < 5

ADVERSE EVENTS:
Time Frame: All AEs were collected from the signature of the informed consent form until the last visit of the subject in the study (up to 22 weeks after the final dose of study treatment) regardless of relationship to study treatment, up to approximately 44 weeks. Any SAE with a start date after the Safety Follow-Up Period was not required to be reported unless the Investigator thought that the event might be related to either the study treatment, study treatment administration, or a protocol procedure
Description: All AEs and SAEs reported below are related to the Safety Population (safety population included all subjects who receive at least 1 dose of study treatment).
  Data for TEAEs were reported below. A Treatment Emergent Adverse Event (TEAE) is defined as an AE that first occurred or worsened in severity after the first dose of the study treatment.
Groups:
- Arm 1: OKZ 64 mg q4w: refers to subjects initially randomized to receive OKZ q4w and relates to AEs reported for this group during the total 24-week study treatment period
- Arm 2: OKZ 64 mg q2w: refers to subjects initially randomized to receive OKZ q2w and relates to AEs reported for this group during the total 24-week study treatment period
- Arm 3: Placebo q2w: refers to subjects initially randomized to receive placebo and relates only to AEs reported for this group during the 16-week treatment period up to re-randomization
- Arm 4: Placebo-OKZ 64 mg q4w: refers to subjects re-randomized to receive OKZ q4w and relates only to AEs reported for this group during the treatment period after re-randomization from Week 16 to Week 24
- Arm 5: Placebo-OKZ 64 mg q2w: refers to subjects re-randomized to receive OKZ q2w and relates only to AEs reported for this group during the treatment period after re-randomization from Week 16 to Week 24
- Arm 6: Any OKZ 64 mg q4w: refers to a combination of the AEs reported for the OKZ 64 mg q4w group and the Placebo-OKZ 64 mg q4w group
- Arm 7: Any OKZ 64 mg q2w: refers to a combination of the AEs reported for the OKZ 64 mg q2w group and the Placebo-OKZ 64 mg q2w group
- Total: refers to AEs reported for all subjects at all visits
Arm/Group | Arm 1: OKZ 64 mg q4w | Arm 2: OKZ 64 mg q2w | Arm 3: Placebo q2w | Arm 4: Placebo-OKZ 64 mg q4w | Arm 5: Placebo-OKZ 64 mg q2w | Arm 6: Any OKZ 64 mg q4w | Arm 7: Any OKZ 64 mg q2w | Total
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/139 | 0/69 | 0/26 | 0/32 | 0/186 | 0/171 | 0/368
Serious Adverse Events (participants affected / at risk) | 6/160 | 12/139 | 0/69 | 0/26 | 0/32 | 6/186 | 12/171 | 18/368
Other Adverse Events (participants affected / at risk) | 38/160 | 38/139 | 16/69 | 2/26 | 8/32 | 40/186 | 46/171 | 98/368
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: OKZ 64 mg q4w (N=160) | Arm 2: OKZ 64 mg q2w (N=139) | Arm 3: Placebo q2w (N=69) | Arm 4: Placebo-OKZ 64 mg q4w (N=26) | Arm 5: Placebo-OKZ 64 mg q2w (N=32) | Arm 6: Any OKZ 64 mg q4w (N=186) | Arm 7: Any OKZ 64 mg q2w (N=171) | Total (N=368)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: OKZ 64 mg q4w (N=160) | Arm 2: OKZ 64 mg q2w (N=139) | Arm 3: Placebo q2w (N=69) | Arm 4: Placebo-OKZ 64 mg q4w (N=26) | Arm 5: Placebo-OKZ 64 mg q2w (N=32) | Arm 6: Any OKZ 64 mg q4w (N=186) | Arm 7: Any OKZ 64 mg q2w (N=171) | Total (N=368)
Nasopharyngitis (Infections and infestations) | 7 (7) | 9 (9) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 10 (10) | 18 (18)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 5 (6) | 4 (4) | 0 (0) | 1 (1) | 6 (6) | 6 (7) | 16 (17)
Latent tuberculosis (Infections and infestations) | 6 (6) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 7 (7) | 6 (6) | 13 (13)
Influenza (Infections and infestations) | 0 (0) | 5 (5) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 10 (10)
Alanine aminotransferase increased (Investigations) | 13 (16) | 10 (13) | 0 (0) | 0 (0) | 1 (1) | 13 (16) | 11 (14) | 24 (30)
Aspartate aminotransferase increased (Investigations) | 8 (9) | 9 (10) | 1 (1) | 0 (0) | 1 (1) | 8 (9) | 10 (11) | 19 (21)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 6 (6) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 8 (8) | 11 (12)
Hypertension (Vascular disorders) | 1 (2) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 2 (3) | 4 (4) | 9 (10)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 8 (8)
Injection site erythema (General disorders) | 7 (13) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 7 (13) | 1 (1) | 8 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related information could be made public available only after Sponsors written permission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT02760433/Prot_SAP_000.pdf